CLINICAL TRIAL: NCT06898021
Title: Diagnostic Performance of 3DStent to Assess Stent Expansion
Brief Title: The 3D Stent Study
Status: Recruiting | Type: Observational
Sponsor: CoreAalst BV (Industry)
Responsible Party: Sponsor
Other Study IDs: CA-1013
Record Dates: First submitted 2025-01-22; First posted 2025-03-27 (Actual); Last update posted 2026-01-12 (Actual); Status verified 2026-01

CONDITIONS: Coronary Artery Disease; Percutaneous Coronary Intervention (PCI)
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing PCI: Patient presenting with chronic or acute coronary syndromes (ACS) with a clinical indication for PCI
  Interventions: Diagnostic Test: 3DStent

INTERVENTIONS:
Diagnostic Test: 3DStent — Coronary interventions will be performed according to the standard of care, which includes IVUS guidance. In patients undergoing stent implantation, a 3DStent image acquisition will be done followed by IVUS.

SUMMARY:
The goal of this observational study is to assess the diagnostic performance of 3D Stent to detect stent under-expansion in patients undergoing percutaneous coronary intervention.

The main question it aims to answer is:

The study hypothesis is that 3DStent technology will offer a comparable assessment of stent expansion compared to intravascular imaging.

ELIGIBILITY:
Inclusion Criteria:

* Patient presenting with chronic or acute coronary syndromes (ACS) with a clinical indication for PCI guided by IVUS.

Exclusion Criteria:

1. Age <18 years
2. Coronary lesions requiring total stent length > 48 mm.
3. Body mass index >35 kg/m2
4. Uncontrolled recurrent ventricular tachycardia
5. Cardiogenic shock
6. Unable to provide written informed consent (IC).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting with chronic or acute coronary syndromes (ACS) and a clinical indication for PCI
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-04-11 (Actual); Primary Completion 2027-11-01 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Diagnostic performance of 3DStent to detect stent underexpansion with intravascular ultrasound imaging (IVUS) as a reference. | Periprocedural timeframe
  Diagnostic performance will be evaluated in terms of sensitivity and specificity. Intravascular Ultrasound (IVUS)-derived minimal stent area (MSA) ≤ 5.5 mm2 will be used to define stent underexpansion.

SECONDARY OUTCOMES:
Agreement on minimal stent area (MSA) between 3DStent and Intravascular Ultrasound (IVUS). | Periprocedural timeframe
  Agreement on minimal stent area (MSA), expressed in mm², between 3DStent and Intravascular Ultrasound (IVUS).
Clinical utility of 3DStent for guiding stent optimisation with Intravascular Ultrasound (IVUS) as a reference. | Periprocedural timeframe
  Clinical utility of 3D stent for guiding stent optimization (i.e. post-dilatation) expressed as a percentage compared with Intravascular Ultrasound (IVUS) as the reference
Feasibility of 3DStent acquisition during the procedure | Periprocedural timeframe
  Feasibility of 3DStent acquisition during the procedure will be assessed based on the technical success rate.
Agreement on stent expansion between 3DStent and IVUS. | Periprocedural timeframe
  Agreement on stent expansion, expressed as a percentage between 3DStent and IVUS.
Impact of lesion location (vessel and segment) on 3DStent diagnostic accuracy. | Periprocedural timeframe
  the impact of the lesion location (location of the vessel and location of the vessel segment) on the diagnostic accuracy of 3D Stent will be assessed.
Agreement on maximal calcium arc as assessed by 3DStent, with IVUS as the reference in cases where 3DStent is acquired pre-PCI. | Periprocedural timeframe
  in cases where 3DStent is also acquired before the PCI procedure, there the agreement on maximal calcium arc will be compared between 3DStent and Intravascular Ultrasound (IVUS).
Impact of calcifications on 3DStent diagnostic accuracy. | Periprocedural timeframe
  Impact of calcifications on 3DStent diagnostic accuracy (measured as mean difference in Minimal Stent Area between 3DStent and IVUS)
Agreement on stent underexpansion and MSA between site and core laboratory. | Periprocedural timeframe
  The assessment of stent underexpansion and minimal stent area will be compared between the results of the site and the results of a core laboratory.
Radiation exposure associated with 3DStent | Periprocedural timeframe
  The dose area product will be measured to assess radiation exposure associated with 3DStent.
Procedural time of the 3DStent workflow | Periprocedural timeframe
  The duration of the 3DStent acquisition workflow from the beginning of the centering until the 3DStent reconstruction appears on the screen, will be measured

CONTACTS AND LOCATIONS:
Overall Officials: Adriaan Wilgenhof, Principal Investigator — Cardiovascular Center Aalst; Carlos Collet, Principal Investigator — CoreAalst BV
Locations (4):
- AZORG Ziekenhuis, Aalst, Belgium
- ICPS, Paris, France
- I.R.C.C.S. Ospedale Galeazzi-Sant'Ambrogio, Milan, Italy
- Hospital Clinic, Barcelona, Spain

IPD SHARING:
Plan to Share IPD: No